CLINICAL TRIAL: NCT06288425
Title: Spatial Transcriptomics in Kidney Transplantation
Acronym: SPACE-KiT
Status: Enrolling by invitation | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Jennifer Li, CPI, Nephrologist and Transplant Physician, Western Sydney Local Health District
Other Study IDs: SPACE-KIT
Record Dates: First submitted 2024-02-03; First posted 2024-03-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Transplant Complication; Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dedicated study samples will be collected at baseline and additional time-points based on the study group. Samples will be sent for processing and biobanking at the Westmead Institute for Medical Research
  Blood sampling: all patients will submit blood samples for extraction of genomic material (eg DNA, RNA), peripheral blood mononuclear cells (PBMC) and plasma/serum.
  Kidney biopsy sample: a dedicated sample of kidney biopsy may be collected for the study with the patient's permission. The core will be split so that half the sample is collected in specialised media for spatial transcriptomics and other molecular/proteinomic studies.
  Additional sampling: Mid-stream urine sample for pellet and supernatant and then stored at -80'c, Faecal sample in dedicated gut microbiome kits and then stored at -80'c. These samples will be biobanked and may be used later for proteinomic or microbiome studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- No rejection, normal biopsy (controls): Normal biopsy - no acute tubular injury (ATI), rejection or any other pathology
  Interventions: Other: Non interventional
- Acute kidney injury without evidence of rejection: Biopsy features of acute tubular injury but no evidence of rejection
  Interventions: Other: Non interventional
- Subclinical Rejection: Biopsy features of injury and inflammation but not meeting current diagnostic criteria for acute or chronic rejection
  Interventions: Other: Non interventional
- Acute rejection: Biopsy features of T-cell mediated, antibody-mediated, or mixed rejection
  Interventions: Other: Non interventional
- Isolated vascular rejection: Biopsy features of inflammation in the blood vessels only
  Interventions: Other: Non interventional
- Isolated glomerulitis: Biopsy features of inflammation in the glomeruli only
  Interventions: Other: Non interventional
- Chronic (active) rejection: Biopsy features of chronic rejection - T-cell, antibody or mixed types
  Interventions: Other: Non interventional
- BK virus associated nephropathy (BKVAN): Biopsy features of SV40 positive staining in tubules to diagnose BKVAN
  Interventions: Other: Non interventional

INTERVENTIONS:
Other: Non interventional — Non interventional. Review of clinical, biopsy (histopathological and molecular) features associated with rejection and non-rejection pathology diagnosis

SUMMARY:
The study is an investigator-led, prospective, longitudinal, observational cohort study.

The central hypothesis for this study is that spatial data will reveal new insights to immune cell function and local interactions within the kidney tissue to better predict important clinical outcomes. Investigators aspire to establish a prospective, longitudinal cohort to improve the diagnosis and management of kidney transplant rejection using precision pathology.

By utilising new spatial technologies, the investigators aim to:

* Derive a spatially resolved transcriptomic signature of kidney transplant rejection subtypes
* Derive accurate transcriptomic signatures aligned with key cell types within the transplant kidney
* Develop refinements to histological kidney rejection diagnostic and scoring classification
* Correlate of spatial and refined biopsy scoring features to clinically important outcomes

DETAILED DESCRIPTION:
Primary outcomes: The correlation of kidney transplant rejection subtypes with transcriptomic, spatial and cell-type features

Secondary outcomes: Correlation of the refined biopsy scoring criteria and transcriptomics signatures with:

1. All cause graft loss
2. Death censored graft loss
3. Treatment resistant rejection
4. Delayed graft function (DGF)
5. Biopsy evidence of borderline rejection based on current Banff scoring system
6. Biopsy proven acute rejection - T-cell mediated (TCMR), antibody-mediated (ABMR), mixed
7. Chronic rejection - acute or inactive
8. Interstitial fibrosis scores (IFTA) on kidney biopsy on any biopsies
9. Chronic transplant glomerulopathy on kidney biopsy on any biopsies
10. Development of BK virus associated nephropathy at any time
11. Recurrent disease (original cause of kidney failure) post transplantation at any time
12. Kidney function with serum creatinine, estimated or measured glomerular filtration rate (GFR)
13. Development of albuminuria
14. Surrogate end-points - eGFR slope and iBOX(TM) score
15. Donor-recipient HLA and non-HLA genomic mismatches
16. Recipient proteinomic expression profile

ELIGIBILITY:
Inclusion Criteria:

All participants included in the study must be age ≥ 18 years old at time of enrolment and

1. able to provide informed consent (interpreter permitted) for enrolment
2. consenting to longitudinal follow up (can withdraw post enrolment)
3. consenting to provide samples for biobanking, including blood, urine, faecal and/or kidney biopsy tissue (collected prospectively, separate to routine care)

Exclusion Criteria:

Patients will be excluded from the study if they are

1. unable (or unwilling) to provide consent, or
2. have life-expectancy less than 6-months, or
3. have received a haematopoietic stem cell transplant in the past 5 years.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney transplant (or kidney-pancreas transplant) recipients consenting to this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Kidney biopsy features | At biopsy or during study follow up following biopsy during study (expected 12-months)
  Based on the pathology subtype at original diagnosis
Kidney biopsy transcriptomic signature | At biopsy - based on collected tissue sample
  Based on bulk and/or spatial transcriptomic experiments
Kidney cell type composition | At biopsy - based on collected tissue sample
  Cell type phenotyping of immune and kidney cell types

SECONDARY OUTCOMES:
All cause graft loss | At biopsy or during study follow up after biopsy (expected average over 60-months)
  Graft loss - death censored and death with functioning graft
Death censored graft loss (DCGL) | At biopsy or during study follow up after biopsy (expected average over 60-months)
  Graft loss - excluding cases of death with functioning graft
Treatment resistant rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Persistent rejection despite additional glucocorticoids and/or upscaling of maintenance immunosuppression
Delayed graft function (DGF) | At biopsy or during study follow up after biopsy (within 7 days of transplantation)
  Need for dialysis within 7 days of transplantation
Biopsy evidence of borderline rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on current Banff scoring system - features of inflammation but not meeting acute rejection criteria
Biopsy proven acute rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on current Banff scoring system - features of acute rejection, , any subtype
Chronic rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on current Banff scoring system with features of chronic rejection, any subtype
Interstitial fibrosis scores (IFTA) | At biopsy or during study follow up after biopsy (expected average 12-months)
  features of interstitial fibrosis scores on the biopsy, with or without concurrent inflammation or tubulitis in the scarred areas on biopsy
BK virus associated nephropathy | At biopsy or during study follow up after biopsy (expected average 12-months)
  biopsy evidence of positive SV40 stain in tubules
Kidney function | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on blood creatinine, eGFR
Albuminuria | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on urine albumin to creatinine ratio
Surrogate end-points | At biopsy or during study follow up after biopsy (expected average 12-months)
  eGFR slow and iBOX score
Donor to recipient mismatches | At biopsy or during study follow up after biopsy (expected average 12-months)
  genomic/molecular level, HLA and non-HLA
Proteinomic signature | At biopsy or during study follow up after biopsy (expected average 12-months)
  mass spectrometry or spatial proteinomic changes between groups

CONTACTS AND LOCATIONS:
Overall Officials: Jen Li, FRACP, Principal Investigator — Westmead Hospital
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No